CLINICAL TRIAL: NCT01897207
Title: Phase I/II Study of Vaccination With Antigen Loaded Dendritic Cells (DCs) in Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Silke Gillessen, Prof. Dr., Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG226_02
Record Dates: First submitted 2013-06-26; First posted 2013-07-11 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Cancer of the Prostate
Keywords: prostate cancer; dendritic cells; vaccination
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dendritic cell application (Experimental)
  Interventions: Biological: Dendritic cell application

INTERVENTIONS:
Biological: Dendritic cell application — S.C. injection of peptide pulsed autologous dendritic cells

SUMMARY:
The main aim of this trial is to assess the response rate, the feasibility and toxicity of the treatment with antigen loaded Dendritic Cell Vaccination in Prostate Cancer patients. Furthermore we want to investigate biological responses by measuring markers of in-vivo and ex-vivo immunomodulation.

DETAILED DESCRIPTION:
Dendritic cell (DC)-based immunotherapy is a promising approach to augment tumor antigen-specific T cell responses in cancer patients. However, tumor escape with down-regulation or complete loss of target antigens may limit the susceptibility of tumor cells to the immune attack. Concomitant generation of T cell responses against several immunodominant antigens may circumvent this potential drawback. In this phase I/II clinical trial, the investigators determined the immunostimulatory capacity of autologous DC pulsed with multiple T cell epitopes derived from four different prostate-specific antigens in patients with advanced hormone-refractory prostate cancer. Autologous DC of HLA-A*0201-positive patients are loaded with antigenic peptides derived from prostate stem cell antigen, prostatic acid phosphatase, prostate-specific membrane antigen, and prostate-specific antigen. A strict quality control concerning the expression of surface markers and the migratory capacity of the DC secured optimal stimulatory capacity. DC were applied intradermally six times at biweekly intervals followed by monthly booster injections. Tolerability and PSA response will be investigated. Antigen-specific immune responses will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven prostatic carcinoma
* proven hormonal resistance: tumor progression after orchiectomy or during treatment with hormonal agents. Patients treated with antiandrogens, such as flutamide (Flucinom) or bicalutamide (Casodex), should have been discontinued the drug 6 weeks prior to the trial entry followed by no tumor response within this 6 weeks
* not amenable to curative therapy
* patients with measurable and non-measurable disease may be included. Bone lesions only are considered to be non-measurable
* two consecutive increases of prostate-specific antigen (PSA) should be documented over a previous reference value (N°1). The first increase in PSA (N°2) should occur a minimum of one week from the reference value and be confirmed (N°3). If this value is less than the previous value, the patient is still eligible if the next PSA(N°4) is found to be higher than the second PSA. Serum levels of prostate-specific antigen must be at least 10 microg/l
* Previous radiotherapy is allowed if it has been stopped 4 weeks or more before the trial treatment and did not involve lesions used to evaluate activity of the trial drugs
* one previous chemotherapy (including Estracyt) is allowed, but the chemotherapy should have been stopped at least 6 weeks before study entry
* age >18 years
* performance status 0,1,2 (ECOG, Appendix I)
* no concurrent therapy with steroids
* no uncontrolled infections
* live expectancy more than 3 months
* Human leukocyte antigen (HLA)-Type has to be HLA*A201
* neutrophile count >1500/microl and thrombocytes >100 000/microl
* creatinine <1.5 of upper normal level
* adequate liver function with bilirubin <2 of upper normal level, alanine aminotransferase (ALAT) and aspartate transamionase (ASAT) < 3 x upper normal level
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient registration/randomization, informed consent must be given according to good clinical practice (GCP), and national/local regulations

Exclusion Criteria:

* serious concomitant disease (cardiac, pulmonary and others)
* brain metastasis
* previous splenectomy or radiotherapy to the spleen
* concurrent therapy with immunosuppressive drugs
* chronic immunosuppression (includes transplantation or HIV-infection) HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) (test required) or any other severe uncontrolled infection other neoplastic diseases except: curatively treated basal cell or squamous cell carcinoma of the skin or relapse free for more than 5 years after curative treatment of a neoplasm
* treatment with other investigational drugs during the last month
* severe autoimmune disease
* chemotherapy, radiotherapy or immunotherapy less than 6 weeks before study entry
* Ejection fraction (measured by echocardiography) < 40%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-11; Primary Completion 2009-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
tolerability and toxicity and feasibility of this regimen | directly after vaccination (within 24 h)
response rate or PSA response in non measurable disease | Change from baseline in serum PSA at 6, 10 and 12 weeks
  The given time frame reflects the minimum of PSA values. From Patients receiving more than 6 DC vaccination every 4 weeks PSA was determined until the end of DC vaccination (longest was one and a half year).
ex-vivo immunomodulation | before vaccination, after 6, 10, 12, and up to 85 weeks
  Peripheral blood mononuclear cells (PBMC) isolation and in-vitro restimulation. Measurement of antigen specific immune responses.

SECONDARY OUTCOMES:
pain relief | Change from baseline in pain relief at 2, 4, 6, 8, 10 and 12 weeks
  Changes in pain intensity will be assessed by summarizing score items 9 and 19 of the European Organisation for Research and Treatment of Cancer (EORTC)quality of life questionnaire (QLQ-C30) quality. Additionally, analgesic consumption will be rated by a pain treatment score (PTS).
Overall survival | From first date of treatment until dead

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cerny, Prof. Dr., Study Chair — Department of Medical Oncology, Cantonal Hospital St. Gallen, Switzerland